CLINICAL TRIAL: NCT05017467
Title: The Effect of Centella Asiatica Cream on Scar Tenderness in Patients Who Underwent Open Carpal Tunnel Release Surgery
Brief Title: The Effect of Centella Asiatica Cream on Scar Tenderness Who Underwent Open Carpal Tunnel Release Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mustafa Balevi,MD (Other Government)
Collaborators: Konya Numune Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Mustafa Balevi,MD, MD., Konya Numune Hospital
Organization: Konya Numune Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.10.4.ISM.4.42.00.14-8271
Record Dates: First submitted 2021-04-10; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: To Prevent Scar Formation for Patients Underwent Surgery
Keywords: carpal tunnel syndrome; centella asiatica; surgery; cosmetic outcome; wound healing
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Centella asiatica extract

STUDY DESIGN:
Intervention Model Description: 280 operated patient with carpal tunnel release surgery.
Who Masked: Participant
Masking Description: 280
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vss (Experimental): Vancouver Scar Scale (VSS) at the one, three and 6 months after surgery
  Interventions: Drug: undefinedCentella Asiatica Extract
- QuickDASH , VAS (Experimental): , Quick Disabilities of Arm Shoulder and Hand functional score (QuickDASH) and Visual Analogue Scale (VAS) test was used to determine overall hand function, activities of daily living, work performance, pain, aesthetics, and satisfaction with hand function
  Interventions: Drug: undefinedCentella Asiatica Extract

INTERVENTIONS:
Drug: undefinedCentella Asiatica Extract — All patients were asked about scar hypertrophy, scar tenderness, and pillar pain.
  The scar assessment was performed using the Vancouver Scar Scale (VSS) at the one, three and 6 months after surgery.
  Patients were asked to complete pre- and postoperative functional evaluations. The VAS score and QuickDASH test was used
  Other Names: centella asiatica extract

SUMMARY:
The centella asiatica cream applied to the wrist after the CTR surgery was found to be beneficial in preventing the scar tenderness in the thenar and hypothenar regions of the hand.

DETAILED DESCRIPTION:
Aim: This study was performed to evaluate the efficacy of centella asiatica extract in a cream preparation for the prevention of scar tenderness formation in patients who underwent conventional open carpal tunnel release surgery.

ELIGIBILITY:
Inclusion Criteria: patient underwent open carpal tunnel release surgery -

Exclusion Criteria:before hand surgery and recurrent carpal tunnel release surgery.

-

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-01-05 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
centella asiatica extrate | 10 years
  treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ali Balevi, Principal Investigator — İstanbul Medipol Üniversity,Medical School
Locations (2):
- Turkey (Türkiye) (2):
  - Mustafa Balevi,MD, Konya, Meram
  - Konya

IPD SHARING:
Plan to Share IPD: No